CLINICAL TRIAL: NCT01641835
Title: Optical Coherence Tomography (OCT) Data Collection Study "S-2012-1 Norm-cc"
Brief Title: Optical Coherence Tomography (OCT) Data Collection Study
Status: Completed | Type: Observational
Sponsor: Heidelberg Engineering GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: S-2012-1 NORM-cc
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Results first posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-09

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Normals: No eye disease.

SUMMARY:
Collect OCT data to evaluate the range and age trend of ocular measurements.

DETAILED DESCRIPTION:
This is a prospective, multi-center study. Ocular history and examination will be conducted on consented subjects to determine further participation in the study. Subjects qualified to continue will undergo imaging of both eyes using the SPECTRALIS OCT.

ELIGIBILITY:
Inclusion Criteria:

* Subject is not an employee of the eye clinic.
* Age ≥18 to 90.
* Able and willing to undergo the test procedures, give consent, and to follow instructions.
* Healthy eye without prior intraocular surgery (except cataract surgery and Lasik) and without clinically significant vitreal, retinal or choroidal diseases, diabetic retinopathy, or disease of the optic nerve.
* Caucasian decent (self-reported).
* Negative history of glaucoma.
* Intraocular pressure ≤21mmHg.
* Best corrected visual acuity ≥0.5.
* Refraction between +6 and -6 diopters and astigmatism ≤ 2 diopters.
* Normal visual field with Glaucoma Hemifield Test and Mean Deviation within normal limits.
* Clinically normal appearance of the optic disc, with normal appearing neuroretinal rim with respect to color and shape. The optic disc is examined ophthalmoscopically and by evaluation of stereo photographs.
* When both eyes are eligible, both eyes enter the study for inter-eye asymmetry; one randomly selected eye will be used for all other measures.

Exclusion Criteria:

* Unreliable visual field. The reliability indices should be used as guide as well as the perimetrist's notes.
* Unusable disc stereo photos.
* Inability to undergo the tests.
* Insufficient quality of Spectralis OCT images (this is not determined until after Spectralis OCT examination, and is an unusual circumstance). Minimum requirements are:

  * Retina completely included in image frame,
  * Quality Score ≥ 20 in the stored ART mean images, and
  * For ONH-R scan: Center position error ≤ 100 μm.
* Note: Inability of a subject to perform one of the two scan patterns or insufficient image quality in one scan pattern does not exclude the subject or eye from the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: No eye disease.
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Balwantray Chauhan, PhD, Principal Investigator — Dalhousie University, Halifax, NS, Canada; Claude Burgoyne, MD, Principal Investigator — Devers Eye Institute, Portland, OR, USA; Christopher Girkin, MD, Principal Investigator — Callahan Eye Foundation Hospital, Birmingham, AL, USA; Christian Mardin, MD, Principal Investigator — Augenklinik des Universitätsklinikums Erlangen, Erlangen, Germany; Alexander Scheuerle, MD, Principal Investigator — Universitätsaugenklinik, Heidelberg, Germany
Locations (1):
- Dalhousie University, Halifax, Nova Scotia, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normals
Started | 303
Completed | 303
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Normals
Number analyzed (Participants) | 303
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 195
  >=65 years | 108
Gender [Count of Participants; unit: Participants]
  Female | 150
  Male | 153
Race/Ethnicity, Customized [Number; unit: participants] — Subjects of Caucasian descent
  participants | 303

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoints
Description: The primary endpoints are the structural measurement values of (1) the ONH, (2) the peri-papillary RNFL, and (3) the macula obtained using the Spectralis OCT and the statistical descriptors such as mean, standard deviation, and distribution percentiles.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: microns
Groups:
- Healthy Volunteers: Healthy eye without prior intraocular surgery (except cataract surgery and Lasik) and without clinically significant vitreal, retinal or choroidal diseases, diabetic retinopathy, or disease of the optic nerve
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 303
microns
  peri-papillary RNFL thickness, 12mm circle scan | 97.2 (9.2)
  peri-papillary RNFL thickness, 14mm circle scan | 83.9 (7.9)
  peri-papillary RNFL thickness, 16mm circle scan | 73.9 (7.0)
  Bruch's Membrane Opening - Minimum Rim Width, glob | 336.1 (51.6)
  Macula parameters have not been analyzed | NA (NA) — Posterior pole volume scans and macula volume scanshave been performed in order to allow future analysis of these data. This analysis was not performed yet and analysis is not planned at the moment.

2. Primary Outcome: Bruch's Membrane Opening - Minimum Rim Area, Global
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: microns^2
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 303
microns^2 | 1339.3 (197.7)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Normals: No adverse events were reported.
Arm/Group | Normals
Serious Adverse Events (participants affected / at risk) | 0/303
Other Adverse Events (participants affected / at risk) | 0/303

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less